CLINICAL TRIAL: NCT02934568
Title: An Open-label, Multi-center Rollover Protocol for Patients Who Have Participated in a Novartis-sponsored Ribociclib (LEE011) Study and Are Continuing to Benefit From Ribociclib as Single Agent or in Combination With Other Investigational Treatments
Brief Title: Ribociclib (LEE011) Rollover Study for Continued Access
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X2X01B
Record Dates: First submitted 2016-10-10; First posted 2016-10-17 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Continued Access to Study Treatment(s), Cancers With a Mass, Bulky Tumor, Nodule, Lump, Advanced Cancer, Advanced Solid Tumors, Advanced Solid Malignancies
Keywords: Ribociclib; LEE011
MeSH Terms: interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LEE011 (Experimental): All patients in all combinations with LEE011 will be entered in one arm.
  Interventions: Drug: LEE011

INTERVENTIONS:
Drug: LEE011 — Single agent LEE011 or in combination with other treatments

SUMMARY:
This study is to allow continued use of ribociclib (LEE011) as single agent or in combination with other investigational treatments in patients benefitting from treatment in an eligible Novartis-sponsored ribociclib (LEE011) study that has reached its primary objective(s) or has been halted for other reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently enrolled in an eligible Novartis-sponsored study and receiving ribociclib (LEE011) as single agent or in combination with other investigational treatment.
2. Patient is currently deriving clinical benefit from the study treatment, as determined by the investigator.

Exclusion Criteria:

1. Patient has been permanently discontinued from ribociclib (LEE011) in the parent protocol for any reason.
2. Patients who do not meet parent protocol criteria to continue study treatment.

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients enrolled and received LEE011 | up to 5 years (study duration)
  Continued access to study treatment as a single agent or in combination with other investigational treatments until patients discontinue study
Length of time receiving study treatment | up to 5 years (study duration)
  Assessed by duration in days from start of study treatment until study treatment discontinuation

SECONDARY OUTCOMES:
Frequency and nature of adverse events (AEs), serious adverse events (SAEs), non-fatal SAEs and liver function assays. | up to 5 years (study duration)
  The data include only AEs that started or worsened during the on-treatment-period, the treatment-emergent AEs.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The Regents of the Uni of Michigan, Ann Arbor, Michigan
  - Broome Oncology, Johnson City, New York
  - St Jude Childrens Research Hospital, Memphis, Tennessee
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Cologne, North Rhine-Westphalia, Germany
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Madrid, Spain
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com